CLINICAL TRIAL: NCT06831734
Title: Special Use-results Surveillance on Use of Alhemo in Patients With Haemophilia A or Haemophilia B Without Inhibitors A Multi-centre, Open-label, Non-interventional Post-marketing Study to Investigate the Long-term Safety and Clinical Parameters of Treatment With Alhemo in Patients With Haemophilia A or Haemophilia B Without Inhibitors in Routine Clinical Practice Conditions in Japan
Brief Title: Post-marketing Surveillance (Special Use-results Surveillance) on Treatment With Alhemo
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7415-7690; U1111-1286-2960 (Other: Universal trial number)
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Haemophilia A, Haemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — concizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Concizumab: Participants with haemophilia A or haemophilia B without inhibitors will be be treated with commercially available Alhemo according to routine clinical practice at the discretion of the treating physician.
  Interventions: Drug: Concizumab

INTERVENTIONS:
Drug: Concizumab — Participants will be treated with commercially available Alhemo according to routine clinical practice at the discretion of the treating physician. Administration will be according to the approved product labelling. The decision to treat a participant with Alhemo is made at the physician's discretion before and independently from this study.
  Other Names: Alhemo

SUMMARY:
The purpose of the study is to investigate the safety and effectiveness of Alhemo in participants under real-world clinical practice in Japan. Total duration of this study is about 6 years. Participants enrolment will be completed in the first 4 years. The observation period of this study will last for about 2 years for each enrolled participant.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* The decision to initiate treatment with commercially available Alhemo has been made by the participant/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the participant in this study.
* Male or female, age above or equal to 12 years at the time of signing informed consent.
* Diagnosis with Haemophilia A (HA) or Haemophilia B (HB).
* Participant who has never been exposed to concizumab or who starts treatment with concizumab within the past 12 weeks at registration.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Treatment with any investigational drug within 30 days prior to baseline (the starting date of Alhemo treatment).
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* A history of hypersensitivity to any ingredients of Alhemo.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants with haemophilia A or haemophilia B without inhibitors will be be treated with commercially available Alhemo according to routine clinical practice at the discretion of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2031-01-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse reaction (AR) | From baseline (week 0) to end of study (week 104)
  Count of adverse reaction.

SECONDARY OUTCOMES:
Number of serious adverse reaction (SAR) | From baseline (week 0) to end of study (week 104)
  Count of serious adverse reaction.
Number of serious adverse event (SAE) | From baseline (week 0) to end of study (week 104)
  Count of serious adverse event.
Number of thromboembolic adverse event (AE) | From baseline (week 0) to end of study (week 104)
  Count of thromboembolic adverse event.
Number of shock/anaphylaxis adverse event (AE) | From baseline (week 0) to end of study (week 104)
  Count of shock/anaphylaxis adverse event.
Number of treated spontaneous and traumatic bleeding episodes | From baseline (week 0) to end of study (week 104)
  Count of treated spontaneous and traumatic bleeding episodes.
Number of treated spontaneous and traumatic target joint bleeding episodes | From baseline (week 0) to end of study (week 104)
  Count of treated spontaneous and traumatic target joint bleeding episodes.
Number of all treatment requiring bleeding episodes | From baseline (week 0) to end of study (week 104)
  Count of all treatment requiring bleeding episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (9):
- Japan (9):
  - Chiba university hospital_Pediatrics, Chiba
  - St. Marianna University School of Medicine Hospital_Pediatrics, Kanagawa
  - Saitama Medical Univ. Hospital Saitama medical center_Department of Transfusion Medicine and Cell Therapy, Kawagoe
  - Nagano red cross hospital_Pediatrics, Nahano
  - Nanbu Medical Center & Children's Medical Center, Okinawa
  - Kansai Medical University Hospital_Pediatrics, Osaka
  - Saitama Medical Univ. Hospital Saitama medical center_Department of Transfusion Medicine and Cell Therapy, Saitama
  - Matsue red cross hospital_Pediatrics, Shimane
  - National Center for Child Health and Development_Hematology, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com